CLINICAL TRIAL: NCT06096207
Title: Deep Brain Stimulation (DBS) Therapy for Treatment Resistant Depression
Brief Title: DBS for Depression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-0209
Record Dates: First submitted 2023-09-18; First posted 2023-10-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
Keywords: TRD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Discontinuation Phase Group 1 (Experimental): Patients will be randomized into two groups for crossover treatment analysis of different parameter settings for six weeks.
  Interventions: Device: Medtronic SenSight Directional DBS lead
- Discontinuation Phase Group 2 (Experimental): Patients will be randomized into two groups for crossover treatment analysis of different parameter settings for six weeks.
  Interventions: Device: Medtronic SenSight Directional DBS lead

INTERVENTIONS:
Device: Medtronic SenSight Directional DBS lead — At the ninth month post DBS implantation, the participant will enter a discontinuation phase of a duration of 6 weeks. The device will be turned on and off without participants' knowledge. After 6 weeks, the device will be turned back on if it was off. Whether the stimulation is active or not, it will be double blinded.

SUMMARY:
The goal of this clinical trial is to demonstrate the feasibility and safety of deep brain stimulation in treatment resistant depression. The main questions it aims to answer are:

* Is deep brain stimulation effective in treating treatment resistant depression?
* Does deep brain stimulation improve overall clinical well-being and functioning?

Participants will be implanted with a deep brain stimulation device. They will then be monitored over a 5-year period by using multiple questionnaires to track their depression symptoms. The device will be turned off at certain time points, unbeknown to the participant, to show the efficacy of the device when it is turned on. The device will be ON for 8.5 months and OFF for 3.5 months during the first year.

Researchers will compare questionnaire scores when the device is off versus on to see if the device is working in reducing depression.

DETAILED DESCRIPTION:
This initial study at Northwell Health has the purpose to demonstrate the feasibility and safety of performing slMFB DBS as a treatment for TRD at Northwell Health as well as more clearly establish efficacy. The investigators hypothesize that DBS targeting can be consistently placed in the supero-lateral branch of the medial forebrain bundle (slMFB) after identification using diffusion tensor imaging and fiber tract analysis, as performed in DBS at UTHealth. The investigators will implant the Medtronic SenSight Directional DBS lead at this target location.

ELIGIBILITY:
Inclusion Criteria:

1. Major Depression Disorder (MDD) or Bipolar Disorder (I /II) diagnosed by Structured Clinical Interview for DSM-V (SCID I/DSM-V)
2. Age 18 - 65 years.
3. 24-item Hamilton Depression Rating Scale (HDRS) score of at least 21 on the first 17 items and/or Montgomery-Asburg Depression Rating Scale (MADRS) score of at least 21.
4. World Health Organization Disability Assessment Scale 2.0(WHODAS2.0) score of 19 or more
5. A recurrent (equal or >4 episodes) or chronic (episode duration equal or higher >2 years) course AND a minimum of 5 years since the onset of the first depressive episode. Major impairment in functioning or potentially severe medical outcomes (repeated hospitalizations, serious suicidal or other self-injurious behavior) over lifetime history as determined by an investigator
6. As determined by the study psychiatrist/investigator, has treatment resistant depression defined as failure to respond to: 6.1. Adequate trials (equal or >6 weeks at an adequate dose) of primary antidepressants from at least 3 different classes AND; 6.2. adequate trials (equal>4 weeks at an adequate dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants,neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant) AND; 6.3 An adequate trial of ECT (>6 bilateral treatments), or inability to tolerate an adequate ECT trial, AND; 6.4 An adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist).
7. Able to comply with the operational and administrative requirements of participation in the study.
8. Able to give written informed consent
9. Major Depressive Disorder (MDD) or Bipolar Disorder (I/II) is the primary psychiatric diagnosis in the medical opinion of an investigator.
10. On a stable psychiatric medication regimen beginning at least 6 weeks prior to enrollment and continuing through the first 6 months of the study, as determined by the investigator. Psychiatric medication changes can be made during the entirety of the subject's study participation but would be limited to the clinical judgment of the PI/study psychiatrist.
11. At enrollment, provides the following information from at least two (2) verifiable contacts who reside within a 10-mile radius of the patient: name, relationship to patient, address (email mail); and telephone (mobile, home, work as applicable).
12. Agrees to allow medical records requests and communications of any type to any and all health care providers who have seen the patient within five years of screening or enrollment.
13. For the duration of study participation, agrees to be followed by a licensed psychiatrist and/or other licensed mental health practitioner on a regularly scheduled basis.
14. FOR AGES 18-21: An average of at least 3 in the following subdomains on the Psychological Maturity Scale (PMS): questions 1-6, "Ego Resilience"; questions 7-13, "Self-Awareness"; questions 14-17, "Autonomy"; questions 18-21, Flexibility".
15. FOR AGES 18-21: Residing with a caretaker or having oversight of a caretaker.

Exclusion Criteria

1. Patients with any lifetime history of psychosis or psychotic disorder, according to DSM-V diagnostic criteria, or in the medical opinion of the PI/study psychiatrist.
2. Any finding on the preoperative magnetic resonance imaging (MRI) scan that, in the opinion of the principal investigator and after consultation with the neuroradiologist, is, or might be, considered clinically significant such that participation in the study: (a) seems likely to increase the medical risk to the subject sufficient to outweigh the potential benefit to study participation; (b) seems likely to jeopardize the subject's ability to complete the study or fulfill all study requirements per protocol; or (c) may impact he integrity of the data or the validity of the results.
3. Any previous surgery to destroy the treatment target (superolateral MFB) rendering it either unilaterally or bilaterally damaged such that it cannot be effectively stimulated, as visualized by pre-operative MRI scans, in the medical opinion of the PI
4. Any surgical contraindications to undergoing DBS, including labeled contraindications for DBS and/orinability to undergo presurgical MRI (cardiac pacemaker, implantable defibrillator or other implantablestimulator, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation, significant cardiac or other medical risk factors for surgery. DBS contraindications include patients who are unable to properly operate the neurostimulator, and patientswho will be exposed to MRI or diathermy. MRI and diathermy (e.g., shortwave diathermy, microwave diathermy or therapeutic ultrasound diathermy) are contraindicated because the energy can be transferred through the implanted System (or any of the separate implanted components), which can cause tissue damage and can result in severe injury or death. Diathermy can damage parts of the neurostimulation system.
5. Refusal of an adequate trial of ECT in the medical opinion of the study psychiatrist or PI following consultation with a study psychiatrist.
6. History of stimulation intolerance in any area of the body.
7. Within six (6) months of the enrollment date, has been diagnosed with, or has met the diagnostic criteria for, a substance abuse disorder (SUD) according to DSM-V criteria.
8. Women of childbearing potential who, at enrollment or during the study: (a)have a positive urine pregnancy test; (b) are heterosexually active without the usage of a medically acceptable, highly effect contraceptive method* (≤1% pregnancy rate); or (c) are planning to become pregnant during the 60-month course of this study, as determined by the PI. *Examples include tubal ligation, vasectomized partner, IUD or IUS (intrauterine device or system), and long-acting reversible contraceptives (LARC).
9. Active suicidal ideation with intent, suicide attempt within the last six months, more than three suicide attempts within the last two years, or serious suicide risk as determined by the study psychiatrists.
10. Participation in another drug, device, or biologics trial within the preceding 30 days
11. Presence of a condition requiring routine MRIs.
12. Presence of a condition requiring diathermy.
13. Subject is on anticoagulant medication.
14. Prior to enrollment or during the course of the study and in the opinion of the PI, has a history of an medical, psychiatric, physical or non-physical disease, disorder, condition, injury, or disability; or has a non-medical reason (e.g., financial, logistical, personal, other) that: (a) may pose a significant risk to the patient; (b) may increase the possibility that the subject is unlikely to successfully complete all of the requirements of the study according to the study protocol; or (c) may adversely impact the integrity of the data or the validity of the study results.
15. Subjects without a fixed home address or stable living situation, in the opinion of the Principal Investigator.
16. Subjects involved in activities involving significant radiation exposure in the past year.
17. Receiving TMS after DBS implantation
18. Any mania or manic episodes within 5 years of enrollment according to DSM-V diagnostic criteria, or in the medical opinion of the PI/study psychiatrist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2030-10-18 (Estimated); Study Completion 2038-10-18 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 12 months
  The MADRS is the Montgomery-Asberg Depression Rating Scale, which at 12 months will be the primary endpoint. The investigators hypothesize is that there will be a significant effect of being stimulated (ON) versus not simulated (OFF) on MADRS scores. Also, that at 12 months 50% of the patients will be responders.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Scale 2.0 (WHODAS2.0) | 12 months
  WHODAS2.0 measures functional impairment. The investigators hypothesize that there will be a significant effect of being stimulated (ON) versus not simulated (OFF) on WHODAS2.0 scores.
Clinical Global Impressions (CGI) rated severity | 12 months
  CGI is a clinician-determined summary based on all available information including severity, global improvement or change, and therapeutic response. The investigators hypothesize that there will be a significant effect of being stimulated (ON) versus not simulated (OFF) on CGI.
Measuring MADRS during discontinuation cross over weeks | 6 weeks
  Depression scores when the device is turned ON verses OFF, as assessed by the MADRS sale. The investigators hypothesize that MADRS values will differ significantly during the two-week period of discontinuation versus the 4-week period of ON.

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Fenoy, MD, Principal Investigator — Northwell Health
Locations (1):
- Zucker Hillside Hospital, Queens, New York, United States

REFERENCES:
- [Background] Fenoy AJ, Schulz P, Selvaraj S, Burrows C, Spiker D, Cao B, Zunta-Soares G, Gajwani P, Quevedo J, Soares J. Deep brain stimulation of the medial forebrain bundle: Distinctive responses in resistant depression. J Affect Disord. 2016 Oct;203:143-151. doi: 10.1016/j.jad.2016.05.064. Epub 2016 Jun 3. PMID 27288959
- [Background] Fenoy AJ, Schulz PE, Selvaraj S, Burrows CL, Zunta-Soares G, Durkin K, Zanotti-Fregonara P, Quevedo J, Soares JC. A longitudinal study on deep brain stimulation of the medial forebrain bundle for treatment-resistant depression. Transl Psychiatry. 2018 Jun 4;8(1):111. doi: 10.1038/s41398-018-0160-4. PMID 29867109
- [Background] Fenoy AJ, Schulz PE, Sanches M, Selvaraj S, Burrows CL, Asir B, Conner CR, Quevedo J, Soares JC. Deep brain stimulation of the "medial forebrain bundle": sustained efficacy of antidepressant effect over years. Mol Psychiatry. 2022 May;27(5):2546-2553. doi: 10.1038/s41380-022-01504-y. Epub 2022 Mar 14. PMID 35288633

DOCUMENTS (1):
  • Informed Consent Form (2025-11-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT06096207/ICF_003.pdf